CLINICAL TRIAL: NCT01320852
Title: PET Scan as a Screening Tool for Liver Transplant in Patients With HCC
Brief Title: PET Scan as a Screening Tool for Liver Transplant in Patients With Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, peter metrakos, Director Multiorgan Transplant Program-MUHC, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: BMD-09-209
Record Dates: First submitted 2010-12-22; First posted 2011-03-23 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Transplant
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Magnetic Resonance Spectroscopy

ARMS (2):
- Milan Criteria (Active Comparator): Patients meeting the Milan Criteria
  Interventions: Other: PET Scan
- No Milan Criteria (Other): Patients not meeting the Milan Criteria
  Interventions: Other: PET Scan

INTERVENTIONS:
Other: PET Scan — All patients will have a PET scan as part of their pre-transplant assessment

SUMMARY:
This study aims at testing the utility of PET Scan as a screening tool for liver transplantation in patients with Hepatocellular Carcinoma. Patients being worked up for liver transplant for hepatocellular carcinoma will undergo a PET Scan and will be followed until 2 years after transplantation. At that time survival data will be analysed according to PET Scan results to determine if it can be used to predict outcome.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient over 18 years of age
* Diagnosis of HCC confirmed by histology if available or by two imaging modalities
* Able to give written informed consent prior to any study specific screening procedures with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.

Exclusion Criteria:

* Unable to give consent to the study
* Unable to undergo a PET Scan

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-12; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Overall Survival | up to death
  The primary objective of the study is to compare, according to PET scan results, the post-transplantation overall survival of patients meeting Milan criteria to those not meeting Milan criteria

CONTACTS AND LOCATIONS:
Locations (1):
- McGill Univeristy Health Centre, Montreal, Quebec, Canada